CLINICAL TRIAL: NCT07180550
Title: Evaluation of the Acute Effects of High-intensity Interval Aerobic Training, Moderate- and High-intensity Functional Training, and Moderate-intensity Functional Training
Brief Title: Acute Effects of High-intensity Interval Aerobic and Functional Training at Different Intensities
Acronym: HIIT-HIFT-FT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European University Miguel de Cervantes (Other)
Collaborators: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PI-DOC008-HIIT-HIFT-FT
Record Dates: First submitted 2025-09-09; First posted 2025-09-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: High Intensity Interval Training (Cycling); High Intensity Interval Training (Running); High Intensity Functional Training; Moderate Intensity Functional Training; High Intensity Traditional Strength Training; Moderate Intensity Traditional Strength Training
Keywords: Metabolic demand; Oxygen consumption; Heart rate variability; Interval training; Strength training
MeSH Terms: interventions — High-Intensity Interval Training; Running

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, crossover interventional study
Who Masked: Investigator
Masking Description: The researcher responsible for analyzing the data will be blinded to the study conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- High-intensity interval training (running) (Experimental): Participants will perform a high-intensity interval training based on six sets of 2-minute runs at an intensity of 90-95% of the maximal aerobic speed (MAS) on a treadmill. The recovery between each set will be 2 minutes, during which the subject will walk at an intensity of 50-60% of MAS.
  Interventions: Other: High-intensity interval training, running
- High-intensity interval training (cycling) (Experimental): Participants will perform a high-intensity interval training based on six sets of 2-minute cycling will be performed at an intensity of 90-95% of the maximal heart rate on a stationary bike. The recovery between each set will be 2 minutes, during which the subject will cycle at an intensity of 50-60% of maximal heart rate.
  Interventions: Other: High-intensity interval training, cycling
- High-intensity functional training (Experimental): Participants will perform a high-intensity functional training based on three sets of six repetitions will be performed at 80% of the one repetition maximum (1-RM) for six exercises. The recovery between exercises will be the minimum time required to switch from one exercise to the next, and between sets, it will be two minutes. Participants will be instructed to move the load as quickly as possible during each repetition.
  Interventions: Other: High-intensity functional training
- Moderate-intensity functional training (Experimental): Participants will perform a moderate-intensity functional training based on three sets of six repetitions will be performed at 60% of the 1-RM for six exercises. The recovery between exercises will be the minimum time required to switch from one exercise to the next, and between sets, it will be two minutes. Participants will be instructed to move the load as quickly as possible during each repetition.
  Interventions: Other: Moderate-intensity functional training
- High-intensity traditional training (Experimental): Participants will perform a high-intensity traditional training based on three sets of six repetitions will be performed at 80% of the 1-RM for six exercises. The recovery after each set will be two minutes of passive rest. Participants will be instructed to move the load as quickly as possible during each repetition.
  Interventions: Other: High intensity traditional strength training
- Moderate-intensity traditional training (Experimental): Participants will perform a high-intensity traditional training based on three sets of six repetitions will be performed at 60% of the 1-RM for six exercises. The recovery after each set will be two minutes of passive rest. Participants will be instructed to move the load as quickly as possible during each repetition.
  Interventions: Other: Moderate intensity traditional strength training

INTERVENTIONS:
Other: High-intensity interval training, running — Six sets of 2-minute runs will be performed at an intensity of 90-95% of the maximal aerobic speed (MAS) on a treadmill. The recovery between each set will be 2 minutes, during which the subject will walk at an intensity of 50-60% of MAS.
  Arms: High-intensity interval training (running)
Other: High-intensity interval training, cycling — Six sets of 2-minute cycling will be performed at an intensity of 90-95% of the maximal heart rate on a stationary bike. The recovery between each set will be 2 minutes, during which the subject will cycle at an intensity of 50-60% of maximal heart rate.
  Arms: High-intensity interval training (cycling)
Other: High-intensity functional training — Three sets of six repetitions will be performed at 80% of the one repetition-maximum (1-RM) for six exercises. The recovery between exercises will be the minimum time required to switch from one exercise to the next, and between sets, it will be two minutes. Participants will be instructed to move the load as quickly as possible during each repetition.
  Arms: High-intensity functional training
Other: Moderate-intensity functional training — Three sets of six repetitions will be performed at 60% of the 1-RM for six exercises. The recovery between exercises will be the minimum time required to switch from one exercise to the next, and between sets, it will be two minutes. Participants will be instructed to move the load as quickly as possible during each repetition.
  Arms: Moderate-intensity functional training
Other: Moderate intensity traditional strength training — Three sets of six repetitions will be performed at 60% of the 1-RM for six exercises. The recovery after each set will be two minutes of passive rest. Participants will be instructed to move the load as quickly as possible during each repetition.
  Arms: Moderate-intensity traditional training
Other: High intensity traditional strength training — Three sets of six repetitions will be performed at 80% of the 1-RM for six exercises. The recovery after each set will be two minutes of passive rest. Participants will be instructed to move the load as quickly as possible during each repetition.
  Arms: High-intensity traditional training

SUMMARY:
Moderate-intensity physical exercise is widely recognized for its health benefits, yet time constraints limit adherence. High-intensity interval training (HIIT) has gained popularity as a more time-efficient alternative, eliciting significant cardiovascular, respiratory, metabolic, and neuromuscular responses. More recently, functional strength exercises have been integrated into high-intensity training, leading to high-intensity functional training (HIFT) and moderate-intensity functional training (MIFT). However, the acute physiological responses to these modalities remain underexplored compared to traditional HIIT (running or cycling) and strength training. This study aims to assess and compare the acute cardiovascular, metabolic, and neuromuscular responses of HIFT, MIFT, HIIT, and traditional strength training in healthy, physically active adults to inform their potential application in special populations.

DETAILED DESCRIPTION:
Moderate-intensity physical exercise has long been a cornerstone in promoting health and well-being. However, despite its well-documented benefits, an exclusive focus on this training modality may overlook some important limitations. One such limitation is the challenge of dedicating sufficient time to physical activity to achieve health and fitness goals. Given this constraint, recent years have witnessed a significant shift in training modalities, moving away from continuous moderate-intensity exercise approaches [e.g., 55-70% of peak heart rate (HRpeak) or 40-60% of maximal oxygen uptake (VO₂max)] toward higher-intensity interval training protocols (e.g., >90% HRpeak or >85% VO₂max), thereby enhancing time efficiency and enjoyment for practitioners.

In this context, the most common type of training is high-intensity interval training (HIIT). HIIT consists of performing brief, high-intensity cyclic and continuous efforts (e.g., running or cycling) separated by predefined rest periods while using a single exercise modality. These short efforts (e.g., 1 to 4 minutes) at high intensity, whether cycling or running, elicit substantial cardiovascular, respiratory, metabolic, and neuromuscular stimuli, which can persist for hours after the workout.

Recently, this training approach has incorporated functional strength exercises-movements that mimic natural movement patterns and have practical applications in daily life-performed at high intensity [e.g., >75% of one-repetition maximum (1RM)] and following a circuit-based exercise organization (i.e., performing one exercise after another rather than using simple sets and pauses), a modality commonly referred to as high-intensity functional training (HIFT). Reducing the intensity of prescribed functional exercises (e.g., 60% 1RM) brings the training program closer to the demands of daily activities, a modality commonly known as moderate-intensity functional training (MIFT). However, both HIFT and MIFT define their intensity theoretically, based on the relative intensity concerning the maximum dynamic concentric strength that individuals can develop in each exercise (%1RM). Meanwhile, the cardiovascular, respiratory, metabolic, and neuromuscular demands of these methodologies remain largely unexplored compared to running-based HIIT (HIIT-R), cycling-based HIIT (HIIT-C), and traditional strength training with moderate (M-FT) and high (H-FT) loads in healthy, physically active adults. Therefore, before these methods can be applied to special populations (e.g., individuals with chronic cardiovascular or respiratory diseases, cancer, or older adults), it is essential to first understand their acute response in healthy, physically active individuals.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older.
* Have at least 6 months of experience in strength training with intensities greater than 75% of one maximum repetition (1-RM).
* Be classified as active according to the International Physical Activity Questionnaire (IPAQ) score.

Exclusion Criteria:

* Musculoskeletal injury within the 6 months prior to the first visit to the laboratory.
* Recent major surgery (<3 months).
* Having a medical condition in which physical activity is contraindicated (assessed with the Physical Activity Readiness Questionnaire, PAR-Q+).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-10-12 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | Week 0 (baseline), Weeks 1-4 (during intervention and 24, 48, and 72 hours post-intervention)
  The heart rate variability (HRV) of the participants will be assessed by monitoring their heart rate, which reflects the variation in the intervals between heartbeats (R-R intervals). This measure is a useful tool in monitoring patient health, as it estimates the balance between the sympathetic and parasympathetic activity of the autonomic nervous system. To evaluate heart rate variability, a Polar H10 heart rate monitor (Polar Electro Oy, Kempele, Finland) and a mobile application, specifically Elite HRV, will be used. Heart rate variability will be monitored daily during the week leading up to the initial assessment visits. Participants will be instructed to take the measurement for the first 5 minutes upon waking and while fasting.
  Subsequently, heart rate variability will be assessed immediately before each training condition, as well as immediately after, at 2, 24, 48, and 72 hours after finishing each training condition.

SECONDARY OUTCOMES:
Post-exercise oxygen debt | Weeks 2-4 (after every intervention session)
  The oxygen debt (EPOC) will be calculated every minute during the 12 minutes following the completion of exercise using the following formula: EPOC (L·min-¹) = oxygen consumption (VO2) post-exercise (L·min-¹) - VO2 at rest (L·min-¹). Subsequently, EPOC will be converted into energy expenditure, using the conversion of 1L of O2 = 4.64 kcal, to exclude the rapid glycolytic resynthesis of adenosine triphosphate (ATP) as part of the conversion of O2 consumption into energy expenditure (EE).
Delayed onset muscle soreness | Weeks 2-4 (24, 48, and 72 hours post-intervention)
  This will be recorded using a visual analog scale, with a score ranging from 0 (no pain) to 10 (worst possible pain), immediately after the exercise and at 24, 48, and 72 hours after completing the training session. To quantify the pain and standardize the measurements, participants will be asked to perform 5 rapid repetitions of sitting down and standing up from a chair, as well as 5 rapid push-up repetitions, after which they will respond to the question, "How sore are your legs/arms?".
Satisfaction with the type of training | Weeks 2-4 (right after every intervention session and 24 hours post-intervention)
  It will be evaluated at the end of each session using a numerical scale from 0 to 10, where the highest score indicates maximum satisfaction with the type of training.
Subjective post-exercise fatigue | Weeks 2-4 (right after every intervention session and 24 hours post-intervention)
  It will be measured using the perceived fatigue scale (ROF). This is a numerical scale that ranges from 0 (no fatigue) to 10 (total fatigue or exhaustion), with five descriptors and five diagrams to help the individual understand the scale and make an assessment. This evaluation will be conducted immediately after the exercise session and 24 hours after completion.
Perceived effort | Weeks 2-4 (right after every intervention session and 24, 48, and 72 hours post-intervention)
  It will be monitored during the six experimental conditions using the Rate of Perceived Exertion (RPE CR-10) scale. The RPE will be recorded after each set or circuit round. Immediately after completing the last set of each condition, participants will be asked to indicate their perceived effort for the entire session. Subsequently, it will be recorded at 24, 48, and 72 hours after the completion of each condition.
Gas exchange analysis | Weeks 2-4 (during intervention sessions)
  The values of mean and peak gas exchange (ml·kg-1·min-1) during the intervention sessions. The gas analyzer that will be used in this study (Cortex Metalyzer 3B, Leipzig, Germany).

OTHER OUTCOMES:
Physical activity levels | Week 0 (baseline)
  The physical activity levels of the participants will be evaluated using the International Physical Activity Questionnaire (IPAQ). This questionnaire consists of 7 questions that will allow for the stratification of physical activity levels.
Cardiorespiratory fitness | Week 1 (baseline)
  The mean and peak values for gas exchange will be recorded in ml/kg·min. The gas analyzer used in this study is the Cortex Metalyzer 3B (Leipzig, Germany). Cardiorespiratory capacity will be determined using a maximum stress test:
  Incremental Ramp Exercise Test on Treadmill (H/P/Cosmos Pulsar, Southern, Germany): The test will begin with a 2-minute warm-up at 7 km/h and a 1% incline. Following this, the test will start at 9 km/h and will increase by 0.5 km/h each minute until exhaustion.
Cardiorespiratory fitness | Week 1 (baseline)
  The mean and peak values for gas exchange will be recorded in ml/kg·min. The gas analyzer used in this study is the Cortex Metalyzer 3B (Leipzig, Germany). Cardiorespiratory capacity will be determined using a maximum stress test:
  Incremental Ramp Exercise Test on Bicycle (Wattbike AtomX, Nottingham, England): The test will begin with a 2-minute warm-up at 100W. After this, the power will increase by 20W each minute until exhaustion, defined as the point at which the participant cannot maintain a cadence of ≥50 revolutions per minute (rpm).
1-RM detection | Week 1 (baseline)
  Each participant will perform the 1-RM test for each exercise, completing the full range of motion with a load approximately equal to 3-RM. The load will be increased by 10 kg if the participant is able to complete the repetition and decreased by 5 kg if they are unable to do so. The test will conclude when the participant is unable to lift a load in two consecutive attempts separated by 2 minutes.
Handgrip strength | Week 0 (baseline)
  Handgrip strength will be assessed using the hand-held Jamar® Plus Smart Dynamometer (Patterson Medical Ltd., Sammons Preston, Nottinghamshire, UK). Manual grip strength will be recorded on both limbs and the dynamometer will be adjusted to hand size prior to testing. The participant's elbow should be in 90° flexion and the forearm fully supported on a table.
Bioimpedance | Week 0 (baseline)
  The NUTRILAB bioimpedance device (AKERN Srl, Florence, Italy) will be used. This non-invasive method measures the body's resistance and reactance of the body to the passage of a low-intensity electric current and enables the determination of various body parameters. Bioimpedance provides accurate data on body composition. Users will be instructed to remove all metal-containing objects and remain in a supine position on a couch during the measurements, with the legs in 45° abduction, the shoulders in 30° abduction relative to the center of the body and the hands in pronation. After cleaning the skin with alcohol, two adhesive electrodes (Biatrodes Akern Srl, Florence, Italy) will be placed on the surface of the right hand and two on the right foot. The measurement results will be given in different unit measures depending on the specific variable assessed.
Muscle thickness | Week 0 (baseline)
  Muscle thickness the vastus lateralis of the dominant side will be measured using a real-time B-mode ultrasound device with a linear transducer. A water-soluble, hypoallergenic transmission gel will be applied to the probe, to serve as a conductive interface between the probe and the participant's skin. Sufficient gel will be used to prevent compression of the muscle by the probe.
Speed-velocity profile | Week 1 (baseline)
  Three intensities will be determined based on the body weight obtained in the first assessment session: weights corresponding to 50% (low load), 75% (medium load), and 100% (high load) of body weight can be selected. To create the speed-velocity profile, three maximum explosive repetitions will be performed in each of the strength exercises at each load percentage, with a three-minute rest between sets.
Weight | Week 1 (baseline)
  Weight will be assess on kilograms (kg)
Height | Week 1 (baseline)
  Height will be assess on centimeters (cm)
Cardiovascular response | Week 1 (baseline)
  The values for minimum, average heart rate (HR) and peak heart rate (HR) will be recorded using a polar H10 chest strap (Polar Electro Oy, Kempele, Finland) during the maximal stress tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Miguel de Cervantes European University, Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No